CLINICAL TRIAL: NCT02363205
Title: Guided Internet-Delivered and Tailored Cognitive Behaviour Therapy for Adolescents With Depression: a Randomized Controlled Trial
Brief Title: Internet-Delivered Cognitive Behaviour Therapy for Adolescent Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/427-31
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention): Weekly check-up
- internet-delivered CBT (Experimental): Tailored Internet-administrated CBT-Treatment
  Interventions: Behavioral: Tailored Internet-administrated CBT-Treatment

INTERVENTIONS:
Behavioral: Tailored Internet-administrated CBT-Treatment — Guided internet-delivered CBT with chat sessions
  Arms: internet-delivered CBT

SUMMARY:
The purpose of this study is to determine whether tailored internet-administrated cognitive behaviour therapy (CBT) is a feasible approach in the treatment of depressive symptoms and comorbid anxiety symptoms.

DETAILED DESCRIPTION:
As above

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 15-19 years old
* Have symptoms of depression, major depression

Exclusion Criteria:

* Suicidal ideation
* Alcohol addiction
* other major primary psychiatric disorder
* Ongoing psychological treatment
* recent (during last 4 weeks) change in psychiatric medication

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory | Baseline, post treatment, 6 months- and 12 months post treatment
  Change from baseline to post treatment, six months and 12 months post treatment.

SECONDARY OUTCOMES:
Beck Anxiety Inventory (BAI) | Baseline, post treatment, 6 months- and 12 months post treatment
  Change from baseline to post treatment, six months and 12 months post treatment.
Social Interaction Anxiety Scale (SIAS) | Baseline, post treatment, 6 months- and 12 months post treatment
  Change from baseline to post treatment, six months and 12 months post treatment.
The General Self-Efficacy Scale (GSE) | Baseline, post treatment, 6 months- and 12 months post treatment
  Change from baseline to post treatment, six months and 12 months post treatment.
Subscale Life activites, WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) | Baseline, post treatment, 6 months- and 12 months post treatment
  Change from baseline to post treatment, six months and 12 months post treatment.
Knowledge of CBT strategies (developed by the research group) | Baseline, post treatment, 6 months- and 12 months post treatment
  Change from baseline to post treatment, six months and 12 months post treatment.
Patient Health Questionnaire (PHQ) | Baseline, post treatment, 6 months- and 12 months post treatment
  Change from baseline to post treatment
The Mood and Feelings Questionnaire (MFQ) | Baseline, post treatment, 6 months- and 12 months post treatment
  Change from baseline to post treatment, six months and 12 months post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, Principal Investigator — Linkoeping University
Locations (1):
- Linköping University, Linköping, Östergotland, Sweden

REFERENCES:
- [Derived] Topooco N, Bylehn S, Dahlstrom Nysater E, Holmlund J, Lindegaard J, Johansson S, Aberg L, Bergman Nordgren L, Zetterqvist M, Andersson G. Evaluating the Efficacy of Internet-Delivered Cognitive Behavioral Therapy Blended With Synchronous Chat Sessions to Treat Adolescent Depression: Randomized Controlled Trial. J Med Internet Res. 2019 Nov 1;21(11):e13393. doi: 10.2196/13393. PMID 31682572